CLINICAL TRIAL: NCT01303081
Title: Financial Incentive Structures for Smoking Cessation: A Pilot Randomized Trial
Brief Title: Pilot Randomized Control Trial of Financial Incentives for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine and Epidemiology , Division of Pulmonary and Critical Care Medicine, Senior Fellow, Center for Bioethics & Leonard Davis Institute of Health Economics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 812287; RC2AG036592 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Work-site; Incentives; Health Behavior; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Health Behavior; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Usual Care (Active Comparator): Participants will be offered free smoking cessation programs, and be provided web-based education regarding the health and economic benefits of smoking cessation. Participants will also have the opportunity to submit weekly reports on their smoking habits. They will be informed that they will receive reimbursements for completing the surveys that are part of the Way To Quit program and for submitting saliva or urine samples at 14 days and 3 months (among those eligible).
  Interventions: Behavioral: Usual Care
- Individual Rewards (Experimental): Same as USUAL CARE arm, plus financial incentive as follows: if participants quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, they will receive a monetary award from the study investigators.
  Interventions: Behavioral: Individual Rewards
- Fixed Deposits (Experimental): Same as USUAL CARE arm, plus financial incentive as follows: participants will have to deposit a certain monetary amount of their own money as an incentive to quit smoking. If they quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, participants will receive their deposit back. If participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Interventions: Behavioral: Fixed Deposits
- Chosen Deposits (Experimental): Same as USUAL CARE, plus financial incentive as follows: participants will choose their deposit amount (XX = chosen deposit); this same amount will be returned upon success (that is, quit smoking by the target quit date, and having this confirmed by cotinine or anabasine tests). If participants do not quit, their money will be used to support future research studies designed to help people stop smoking. The default deposit will be set to a certain monetary amount for consistency with other arms, and participants can increase or decrease this amount until they reach the amount they want to deposit.
  Interventions: Behavioral: Chosen Deposits
- Competitive Deposits (Pari-Mutuel) (Experimental): Same as USUAL CARE, plus financial incentive as follows: groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. Participants will deposit a certain monetary amount (Y) in an account, and the payout for quitting on this arm will be Y x 6/Q , where Q is the number of quits in the cohort. Again, success will be confirmed by cotinine or anabasine tests, and if participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Interventions: Behavioral: Competitive Deposits (Pari-Mutuel)

INTERVENTIONS:
Behavioral: Individual Rewards — If participants quit smoking by their target quit date, and that is confirmed by cotinine/anabasine tests, they will receive a monetary award from the study investigators.
  Arms: Individual Rewards
Behavioral: Fixed Deposits — Participants will have to deposit a certain monetary amount of their own money as an incentive to quit smoking. If they quit smoking by their target quit date, and that is confirmed by cotinine/anabasine tests, participants will receive their deposit back. If participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Arms: Fixed Deposits
Behavioral: Chosen Deposits — Participants will choose their deposit amount (XX = chosen deposit); this same amount will be returned upon success (that is, quit smoking by the target quit date, and having this confirmed by cotinine/anabasine tests). If participants do not quit, their money will be used to support future research studies designed to help people stop smoking. The default deposit will be set to a certain monetary amount for consistency with other arms, and participants can increase or decrease this amount until they reach the amount they want to deposit.
  Arms: Chosen Deposits
Behavioral: Competitive Deposits (Pari-Mutuel) — Groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. Participants will deposit a certain monetary amount (Y) in an account, and the payout for quitting on this arm will be Y x 6/Q , where Q is the number of quits in the cohort. Again, success will be confirmed by cotinine or anabasine tests, and if participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Arms: Competitive Deposits (Pari-Mutuel)
Behavioral: Usual Care — Participants will receive reimbursements for completing the surveys that are part of the Way To Quit program and for submitting saliva or urine samples at 14 days and 3 months (among those eligible).
  Arms: Usual Care

SUMMARY:
Financial incentives may be more effective than other approaches to smoking cessation, but research is needed to identify the optimal structures of incentives. The investigators will conduct a pilot randomized trial comparing different incentive structures for smoking cessation. Collaborating with Walgreens leadership, the investigators will enroll their employees in this RCT using the investigators new web-based research infrastructure (called the Way to Health platform, and approved as a Prime protocol by the IRB as reference # 811860).

Hypothesis: providing patients with financial incentives can promote healthier behaviors (e.g.: quit smoking).

DETAILED DESCRIPTION:
This study is designed to explore the potential efficacy of using internet-based incentive programs to promote smoking cessation. We also hope to document that we can recruit participants through a web site, as well as investigate what forms of incentives show the most promise. We seek to achieve three specific objectives: (1) assess our ability to recruit participants for several different types of intervention-based smoking programs; (2) document the feasibility of using the internet to accrue and disburse incentive payments; (3) obtain preliminary assessments of which incentive structures show the most promise for future study.

Potential participants will be directed to the Way to Health research portal and will be assessed for eligibility. The web application will automatically verify eligibility based on the results of the survey. If a person is deemed eligible, he or she will be invited to consent to participate in a non-pharmacologic smoking cessation study lasting 3 months. Participants who consent will be randomized automatically to one of the 5 intervention arms (including the no-incentive arm) by the web application.

Once the participant consents and submits the necessary financial information, he will gain access to the participant interface. At this point, they will receive detailed descriptions of their assigned incentive structures (or usual care provisions), will indicate their acceptance of their assigned structure and, for those in arms 3, 4, or 5, make their required deposits. Also, he will be prompted to take an initial survey on his baseline smoking habits. The participant will be able to log into this interface at anytime and see a graph of his self-reported smoking habits along with a graph of approximately how much money he has saved compared to his baseline smoking levels. Participants will indicate their preferred method of contact: email, text-messaging, or both. Every week the participant will receive an email or text-message reminder to log in and complete a weekly smoking report. Participants can also log in at any time and report on their smoking habits for a given day or days to improve accuracy. After three months all subjects will be e-mailed to prompt them to log into the web application to take a final smoking habits survey. Participants who report having remained smoke free for the last month of the study will submit saliva (or urine, for participants using any form of nicotine replacement therapy) samples to test for cotinine (or anabasine) to verify that they have quit. Once this has been verified, the participant will be sent whatever financial incentives he has earned and any deposit will be returned.

The design of this study differs from a traditional RCT in two important ways. First, because the goal of this RCT is to focus on mechanisms of behavior change, we include a primary per-protocol analysis designed to determine incentive structures' efficacy by analyzing only participants who accept their assigned incentive structure at the time of randomization. In this analysis, the randomization arm will be entered into the analytic model as an instrumental variable to mitigate potential selection bias. As in a traditional RCT, we will also analyze each incentive structures' effectiveness using an intention-to-treat analysis that includes all randomized participants, regardless of whether they accept the randomly assigned arm. The second difference is that because acceptance rates of the different structures may differ (as we will test in Aim II), we will adapt the probabilities of being randomized to each arm on a weekly basis during the enrollment period to achieve the target numbers of participants in the per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker of 5 cigarettes per day for at least 6 months
* At least 18 years old
* Interested in quitting smoking
* Current full-time employee of Walgreens

Exclusion Criteria:

* Plan to stop working at Walgreens in the next 12 months
* Currently use a form of tobacco other than cigarettes (as this may influence biochemical testing)
* Are unable or unwilling to access the internet
* Are unable to provide informed consent
* Do not have reliable computer or internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Salivary cotinine or urinary anabasine testing (metabolites of nicotine) | at 3 months following the patient-selected target quit date
  The primary measure of smoking cessation will be prolonged abstinence for 3 months, which will be measured by salivary cotinine testing or by urinary anabasine testing (for those participants using nicotine replacement therapy). Saliva samples will be analyzed using semi-quantitative immunochromatographic assay test strips at the University of Pennsylvania. Urine samples will be analyzed using gas chromatography at the Associated Regional and University Pathologists (ARUP) Lab, at the University of Utah.

SECONDARY OUTCOMES:
Salivary cotinine or urinary anabasine testing (metabolites of nicotine) | at 14 days following the patient-selected target quit date
  The secondary measure of smoking cessation will be point-prevalent quit rates at 14 days, which will also be measured by salivary cotinine testing or by urinary anabasine testing (for those participants using nicotine replacement therapy). Saliva samples will be analyzed using semi-quantitative immunochromatographic assay test strips at the University of Pennsylvania. Urine samples will be analyzed using gas chromatography at the Associated Regional and University Pathologists (ARUP) Lab, at the University of Utah.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Halpern, MD, Ph.D., Principal Investigator — University of Pennsylvania, Department of Medicine, Pulmonary, Allergy and Critical Care; Kevin Volpp, MD, Ph.D., Principal Investigator — University of Pennsylvania; Benjamin French, MS, Ph.D., Principal Investigator — University of Pennsylvania; Dylan Small, Ph.D., Principal Investigator — University of Pennsylvania; David Asch, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Halpern SD, Madison KM, Volpp KG. Patients as mercenaries?: the ethics of using financial incentives in the war on unhealthy behaviors. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):514-6. doi: 10.1161/CIRCOUTCOMES.109.871855. No abstract available. PMID 20031885
- [Background] Volpp KG, Pauly MV, Loewenstein G, Bangsberg D. P4P4P: an agenda for research on pay-for-performance for patients. Health Aff (Millwood). 2009 Jan-Feb;28(1):206-14. doi: 10.1377/hlthaff.28.1.206. PMID 19124872
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Lussier JP, Heil SH, Mongeon JA, Badger GJ, Higgins ST. A meta-analysis of voucher-based reinforcement therapy for substance use disorders. Addiction. 2006 Feb;101(2):192-203. doi: 10.1111/j.1360-0443.2006.01311.x. PMID 16445548
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] Hughes JR. Motivating and helping smokers to stop smoking. J Gen Intern Med. 2003 Dec;18(12):1053-7. doi: 10.1111/j.1525-1497.2003.20640.x. PMID 14687265
- [Background] Hennrikus DJ, Jeffery RW, Lando HA, Murray DM, Brelje K, Davidann B, Baxter JS, Thai D, Vessey J, Liu J. The SUCCESS project: the effect of program format and incentives on participation and cessation in worksite smoking cessation programs. Am J Public Health. 2002 Feb;92(2):274-9. doi: 10.2105/ajph.92.2.274. PMID 11818305
- [Background] Donatelle R, Hudson D, Dobie S, Goodall A, Hunsberger M, Oswald K. Incentives in smoking cessation: status of the field and implications for research and practice with pregnant smokers. Nicotine Tob Res. 2004 Apr;6 Suppl 2:S163-79. doi: 10.1080/14622200410001669196. PMID 15203819
- [Background] Volpp KG, Gurmankin Levy A, Asch DA, Berlin JA, Murphy JJ, Gomez A, Sox H, Zhu J, Lerman C. A randomized controlled trial of financial incentives for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):12-8. doi: 10.1158/1055-9965.EPI-05-0314. PMID 16434580
- [Background] Coffield AB, Maciosek MV, McGinnis JM, Harris JR, Caldwell MB, Teutsch SM, Atkins D, Richland JH, Haddix A. Priorities among recommended clinical preventive services. Am J Prev Med. 2001 Jul;21(1):1-9. doi: 10.1016/s0749-3797(01)00308-7. PMID 11418251
- [Background] Cromwell J, Bartosch WJ, Fiore MC, Hasselblad V, Baker T. Cost-effectiveness of the clinical practice recommendations in the AHCPR guideline for smoking cessation. Agency for Health Care Policy and Research. JAMA. 1997 Dec 3;278(21):1759-66. PMID 9388153
- [Background] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Asch DA. Empirical assessment of whether moderate payments are undue or unjust inducements for participation in clinical trials. Arch Intern Med. 2004 Apr 12;164(7):801-3. doi: 10.1001/archinte.164.7.801. PMID 15078651
- [Background] Halpern SD, Raz A, Kohn R, Rey M, Asch DA, Reese P. Regulated payments for living kidney donation: an empirical assessment of the ethical concerns. Ann Intern Med. 2010 Mar 16;152(6):358-65. doi: 10.7326/0003-4819-152-6-201003160-00005. PMID 20231566
- [Background] Audrain J, Boyd NR, Roth J, Main D, Caporaso NF, Lerman C. Genetic susceptibility testing in smoking-cessation treatment: one-year outcomes of a randomized trial. Addict Behav. 1997 Nov-Dec;22(6):741-51. doi: 10.1016/s0306-4603(97)00060-9. PMID 9426791
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Pomerleau CS, Carton SM, Lutzke ML, Flessland KA, Pomerleau OF. Reliability of the Fagerstrom Tolerance Questionnaire and the Fagerstrom Test for Nicotine Dependence. Addict Behav. 1994 Jan-Feb;19(1):33-9. doi: 10.1016/0306-4603(94)90049-3. PMID 8197891
- [Background] Hymowitz N, Cummings KM, Hyland A, Lynn WR, Pechacek TF, Hartwell TD. Predictors of smoking cessation in a cohort of adult smokers followed for five years. Tob Control. 1997;6 Suppl 2(Suppl 2):S57-62. doi: 10.1136/tc.6.suppl_2.s57. PMID 9583654
- [Background] Kenford SL, Fiore MC, Jorenby DE, Smith SS, Wetter D, Baker TB. Predicting smoking cessation. Who will quit with and without the nicotine patch. JAMA. 1994 Feb 23;271(8):589-94. doi: 10.1001/jama.271.8.589. PMID 8301790
- [Background] Giuffrida A, Torgerson DJ. Should we pay the patient? Review of financial incentives to enhance patient compliance. BMJ. 1997 Sep 20;315(7110):703-7. doi: 10.1136/bmj.315.7110.703. PMID 9314754
- [Background] Delmonico FL, Arnold R, Scheper-Hughes N, Siminoff LA, Kahn J, Youngner SJ. Ethical incentives--not payment--for organ donation. N Engl J Med. 2002 Jun 20;346(25):2002-5. doi: 10.1056/NEJMsb013216. No abstract available. PMID 12075064
- [Background] Dickert N, Grady C. What's the price of a research subject? Approaches to payment for research participation. N Engl J Med. 1999 Jul 15;341(3):198-203. doi: 10.1056/NEJM199907153410312. No abstract available. PMID 10403861
- [Background] Macklin R. On paying money to research subjects: 'due' and 'undue' inducements. IRB. 1981 May;3(5):1-6. No abstract available. PMID 11649367
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Brownson RC, Eriksen MP, Davis RM, Warner KE. Environmental tobacco smoke: health effects and policies to reduce exposure. Annu Rev Public Health. 1997;18:163-85. doi: 10.1146/annurev.publhealth.18.1.163. PMID 9143716
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Rodgers K, Cuevas J, Wileyto EP. Young adult smoking: what factors differentiate ex-smokers, smoking cessation treatment seekers and nontreatment seekers? Addict Behav. 2009 Dec;34(12):1036-41. doi: 10.1016/j.addbeh.2009.06.012. Epub 2009 Jul 5. PMID 19619948
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Cuevas J, Rodgers K, Wileyto EP. Does delay discounting play an etiological role in smoking or is it a consequence of smoking? Drug Alcohol Depend. 2009 Aug 1;103(3):99-106. doi: 10.1016/j.drugalcdep.2008.12.019. Epub 2009 May 14. PMID 19443136
- [Background] Bickel WK, Odum AL, Madden GJ. Impulsivity and cigarette smoking: delay discounting in current, never, and ex-smokers. Psychopharmacology (Berl). 1999 Oct;146(4):447-54. doi: 10.1007/pl00005490. PMID 10550495
- [Background] Johnson MW, Bickel WK, Baker F. Moderate drug use and delay discounting: a comparison of heavy, light, and never smokers. Exp Clin Psychopharmacol. 2007 Apr;15(2):187-94. doi: 10.1037/1064-1297.15.2.187. PMID 17469942
- [Background] Kirby KN, Petry NM, Bickel WK. Heroin addicts have higher discount rates for delayed rewards than non-drug-using controls. J Exp Psychol Gen. 1999 Mar;128(1):78-87. doi: 10.1037//0096-3445.128.1.78. PMID 10100392
- [Background] Baker F, Johnson MW, Bickel WK. Delay discounting in current and never-before cigarette smokers: similarities and differences across commodity, sign, and magnitude. J Abnorm Psychol. 2003 Aug;112(3):382-92. doi: 10.1037/0021-843x.112.3.382. PMID 12943017
- [Background] Jacob P 3rd, Wilson M, Benowitz NL. Improved gas chromatographic method for the determination of nicotine and cotinine in biologic fluids. J Chromatogr. 1981 Jan 2;222(1):61-70. doi: 10.1016/s0378-4347(00)81033-6. PMID 6783675
- [Background] Jacob P 3rd, Yu L, Wilson M, Benowitz NL. Selected ion monitoring method for determination of nicotine, cotinine and deuterium-labeled analogs: absence of an isotope effect in the clearance of (S)-nicotine-3',3'-d2 in humans. Biol Mass Spectrom. 1991 May;20(5):247-52. doi: 10.1002/bms.1200200503. PMID 1883864
- [Background] Greenland S, Schwartzbaum JA, Finkle WD. Problems due to small samples and sparse data in conditional logistic regression analysis. Am J Epidemiol. 2000 Mar 1;151(5):531-9. doi: 10.1093/oxfordjournals.aje.a010240. PMID 10707923
- [Background] Higgins ST, Heil SH, Dantona R, Donham R, Matthews M, Badger GJ. Effects of varying the monetary value of voucher-based incentives on abstinence achieved during and following treatment among cocaine-dependent outpatients. Addiction. 2007 Feb;102(2):271-81. doi: 10.1111/j.1360-0443.2006.01664.x. PMID 17222282
- [Background] Centers for Disease Control and Prevention (CDC). State-specific smoking-attributable mortality and years of potential life lost--United States, 2000-2004. MMWR Morb Mortal Wkly Rep. 2009 Jan 23;58(2):29-33. PMID 19165137
- [Background] Hatsukami DK, Stead LF, Gupta PC. Tobacco addiction. Lancet. 2008 Jun 14;371(9629):2027-38. doi: 10.1016/S0140-6736(08)60871-5. PMID 18555914
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults and trends in smoking cessation - United States, 2008. MMWR Morb Mortal Wkly Rep. 2009 Nov 13;58(44):1227-32. PMID 19910909
- [Background] Donatelle RJ, Prows SL, Champeau D, Hudson D. Randomised controlled trial using social support and financial incentives for high risk pregnant smokers: significant other supporter (SOS) program. Tob Control. 2000;9 Suppl 3(Suppl 3):III67-9. doi: 10.1136/tc.9.suppl_3.iii67. No abstract available. PMID 10982912
- [Background] Prochaska JO, DiClemente CC, Velicer WF, Rossi JS. Standardized, individualized, interactive, and personalized self-help programs for smoking cessation. Health Psychol. 1993 Sep;12(5):399-405. doi: 10.1037//0278-6133.12.5.399. PMID 8223364